CLINICAL TRIAL: NCT03421314
Title: Effect of Zinc and Selenium Supplementation on Clinical and Immunological Parameters on HIV+ Individuals on Antiretroviral Treatment.
Brief Title: Effect of Zinc and Selenium Supplementation on HIV+ Individuals on Antiretroviral Treatment.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Gustavo Reyes-Teran, Principal Investigator, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: C21-16
Record Dates: First submitted 2018-01-10; First posted 2018-02-05 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: HIV; ART; Zinc Deficiency; Selenium Deficiency; Metabolic Complication; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Zinc (Experimental): Participants in this arm will take a daily 30 mg dose of zinc gluconate during 6 months
  Interventions: Dietary Supplement: Zinc gluconate and/or Selenium yeast
- Selenium (Experimental): Participants in this arm will take a daily 200 mcg of selenium yeast during 6 months
  Interventions: Dietary Supplement: Zinc gluconate and/or Selenium yeast
- Zinc + Selenium (Experimental): Participants in this arm will take a daily 30 mg dose of zinc gluconate + 200 mcg of selenium yeast during 6 months
  Interventions: Dietary Supplement: Zinc gluconate and/or Selenium yeast
- Control (No Intervention): Participants in this arm will not take supplementation as a control.

INTERVENTIONS:
Dietary Supplement: Zinc gluconate and/or Selenium yeast — 30 mg dose of zinc gluconate and/or 200 mcg of selenium yeast
  Arms: Selenium; Zinc; Zinc + Selenium

SUMMARY:
The aim of this study is to evaluate the effect of zinc gluconate and/or selenium yeast supplementation during six months on clinical (glucose, cholesterol, triglycerides, bone mineral density and body composition) and immunological (oxidative stress, CD4+ count and pro-inflammatory cytokines) parameters in a population with HIV diagnosis on antiretroviral treatment.

DETAILED DESCRIPTION:
HIV-infected individuals on antiretroviral treatment have lowest risk of AIDS events and more life expectancy. However, antiretroviral treatment does not fully restore the immune system in all individuals due to persistent immune activation and inflammation, increasing the risk of non-AIDS complications, such as insulin resistance, diabetes, hypertension, dyslipidemia, obesity, low bone mass density, oxidative stress and micronutrient deficiencies. Several studies showed that HIV+ patients present zinc and selenium deficiency. Those micronutrients are involved in the pathogenesis of metabolic complications and have a major role in maintaining immune system function. It remains unknown the effect of zinc and selenium supplementation on metabolic and immunological parameters associated to non-AIDS complications.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* >200 CD4+ cells/mL
* >2 years under antiretroviral treatment
* >2 years under virology control (HIV RNA <40 copies/mL)

Exclusion Criteria:

* Patients with opportunistic infection
* Patients taking vitamin-mineral supplements
* Patients with moderate or high cardiovascular risk (Framingham score higher than 10%) and cholesterol LDL >190 mg/dL or triglycerides >500 mg/dL.
* Patients with diabetes or hypertension diagnosis.
* Patients taking drugs for diabetes, hypertension, dyslipidemia or low bone mass density.
* Low adherence to supplementation.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 37 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in zinc and selenium plasmatic levels | Baseline and 24 weeks
  We evaluated the effects of zinc (30mg/d) and selenium (200μg/d) supplementation on plasma zinc and selenium levels.

SECONDARY OUTCOMES:
Counts of CD4+ T cells | Baseline,12 and 24 weeks
Changes in fasting serum glucose | Baseline,12 and 24 weeks
Changes in blood pressure | Baseline,12 and 24 weeks
Changes in lipid peroxidation | Baseline and 24 weeks
  Measure by TBARS
Changes in proinflammatory cytokine profile | Baseline and 24 weeks
  Measure by LUMINEX
Changes in bone metabolism biomarkers | Baseline and 24 weeks
  Changes in osteoprotegerin and RANKL levels
Frequency of CD4+ T cells | Baseline,12 and 24 weeks
  Measure by flow cytometry
Changes in total cholesterol | Baseline,12 and 24 weeks
  in mg/dL
Changes in LDL cholesterol | Baseline,12 and 24 weeks
  in mg/dL
Changes in HDL cholesterol | Baseline,12 and 24 weeks
  in mg/dL
Changes in triglycerides | Baseline,12 and 24 weeks
  in mg/dL
Changes in body weight | Baseline,12 and 24 weeks
  in Kg
Changes in fat mass | Baseline,12 and 24 weeks
  in Kg
Changes in lean soft tissue | Baseline,12 and 24 weeks
  in Kg
Changes in and bone mineral density | Baseline,12 and 24 weeks
  g/cm3

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Reyes Teran, MD, Principal Investigator — Principal investgator
Locations (1):
- Centro de Investigaciones en Enfermedades Infecciosas, Mexico City, Mexico City, Mexico